CLINICAL TRIAL: NCT00540007
Title: A Phase II Multicenter Study of Lenalidomide in Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Lenalidomide in Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0233 / 201104227
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin Lymphoma; Lenalidomide; Anti-neoplastic agents; Thalidomide
MeSH Terms: conditions — Hodgkin Disease | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Lenalidomide daily on days 1-21 (Experimental): * The first group of participants will be assigned to Cohort 1 and if no unacceptable toxicities occur in Cohort 1 then the second group of participants will be assigned to Cohort 2
  * Lenalidomide 25 mg per day PO daily on days 1-21 of a 28 day cycle.
  Interventions: Drug: Lenalidomide
- Cohort 2 - Lenalidomide daily on days 1-28 (Experimental): * The first group of participants will be assigned to Cohort 1 and if no unacceptable toxicities occur in Cohort 1 then the second group of participants will be assigned to Cohort 2
  * Lenalidomide 25 mg per day PO daily on days 1-28 of a 28 day cycle.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid; CC-5013

SUMMARY:
The purpose of this study is to determine the efficacy of lenalidomide in the treatment of relapsed or refractory classic Hodgkin lymphoma(cHL).

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL), an uncommon but significant subtype of lymphoma, is divided into classical HL (cHL) and nodular lymphocyte predominant HL (NLPHL). Progress has been made in cHL therapy resulting in 5-year failure free survival rates between 61%-89% even in the setting of advanced stage or bulky disease. Patients who relapse however, have a variable prognosis ranging from a 8-year overall survival rate of less than 8% for patients who never achieve a remission to 54% for patients with a complete remission lasting greater than 12 months. High dose chemotherapy with autologous stem cell support is the standard of care for patients with relapsed cHL but for those that relapse despite aggressive salvage therapy 20 - 50%, with median remission durations of approximately 6 months. Furthermore, a subset of relapsed HL patients may not be candidates for aggressive salvage regimens. These novel salvage therapies are needed for relapsed/refractory cHL, especially agents without serious late toxicities are particularly attractive in this disease. Advances in the understanding of HL pathogenesis and lenalidomide's mechanisms of action provide substantial rationale for evaluating lenalidomide in HL patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented classical Hodgkin lymphoma that is recurrent or refractory to standard chemotherapy.
* Patients must have relapsed or progressed after at least one prior systemic cytotoxic chemotherapy; prior autologous or allogeneic stem cell transplantation is allowed.
* Measurable disease must be present either on physical examination or imaging studies (CT, MRI, PET/CT). Any tumor mass greater or equal to 1 cm is acceptable.
* Age > 18 years old.
* ECOG performance status of less than or equal to 2 at study entry
* Adequate hematologic, renal, hepatic function as defined by:

  * Absolute neutrophil count greater than or equal to 1000 / uL
  * Platelets greater than or equal to 50,000 / uL
  * Serum creatinine less than or equal to 1.5X institution upper limit of normal (ULN)
  * Total bilirubin less than or equal to 2.0 mg/dL
  * AST (SGOT) and ALT (SGPT) less than or equal to 3 x ULN (if not attributed to cHL)
* Disease free of prior malignancies for greater than or equal to 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements
* Females of childbearing potential (FCBP)† must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* FCBP must have two negative serum or urine pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. The subject may not receive study drug until the Investigator has verified that the results of these pregnancy tests are negative.
* Men must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
* All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist.

Exclusion Criteria:

* Patients who are candidates for high dose chemotherapy and stem cell transplantation and have not yet undergone stem cell transplantation should not be enrolled.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any condition, including the presence of laboratory abnormalities.
* Use of any other anti-cancer drug or therapy, including experimental, within 30 days of enrollment.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Known positive for HIV or infectious hepatitis, type A, B or C.
* Pregnant or breastfeeding females.
* Concurrent use of other anti-cancer agents or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-09-06 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Fehniger, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Wake Forest University Medical School, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett JB, Dredge K, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. Nat Rev Cancer. 2004 Apr;4(4):314-22. doi: 10.1038/nrc1323. No abstract available. PMID 15057291
- [Derived] Fehniger TA, Larson S, Trinkaus K, Siegel MJ, Cashen AF, Blum KA, Fenske TS, Hurd DD, Goy A, Schneider SE, Keppel CR, Wagner-Johnston ND, Carson KR, Bartlett NL. A phase 2 multicenter study of lenalidomide in relapsed or refractory classical Hodgkin lymphoma. Blood. 2011 Nov 10;118(19):5119-25. doi: 10.1182/blood-2011-07-362475. Epub 2011 Sep 21. PMID 21937701
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Started | 38 | 42
Completed | 38 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28 | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Median (Full Range); unit: years] | 34 [25 to 63] | 38 [19 to 84] | 36 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 16 | 24 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Objective Overall Response Rate (ORR) in Relapsed or Refractory cHL.
Description: * Overall response rate = CR + PR
  * Definitions per 2007 Cheson Lymphoma Response Criteria
Time Frame: Through 3.5 years from study entry or until disease progression
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 42
percentage of participants | 21.0 [9.6 to 37.3] | 28.6 [15.7 to 44.6]

2. Secondary Outcome: Safety and Tolerability of Lenalidomide Therapy as Measured by the Number of Participants Who Experience Each Adverse Event (Grade 3 or 4 Adverse Events Only) Refractory cHL.
Description: * Adverse events were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
  * The higher the grade the worse the adverse event was considered
Time Frame: 30 days following the completion of treatment
Measure: Number; unit: participants
Groups:
- Cohort 2: Lenalidomide 25 mg per day PO daily on days 1-28 of a 28 day cycle.
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2
Number analyzed (Participants) | 38 | 42
participants
  Neutropenia | 18 | 20
  Leukopenia | 11 | 13
  Anemia | 10 | 4
  Lymphopenia | 9 | 10
  Thrombocytopenia | 7 | 8
  Fatigue | 3 | 2
  AST | 3 | 1
  ALT | 2 | 1
  Bilirubin | 2 | 2
  Sensory neuropathy | 2 | 0
  Dehydration | 2 | 0
  Infection without neutropenia | 2 | 3
  Infection with neutropenia | 1 | 0
  Edema | 1 | 0
  Dyspnea | 1 | 0
  Pleural effusion | 1 | 0
  Alkaline phosphatase | 1 | 0
  Abdominal pain | 1 | 0
  Low potassium | 3 | 3
  Low sodium | 2 | 2
  Low albumin | 1 | 0
  Low calcium | 1 | 0
  High calcium | 1 | 0
  Low phosphorus | 1 | 0
  Hearing loss | 0 | 1
  Thrombosis/embolism | 0 | 1
  Rash | 0 | 1
  Febrile neutropenia | 1 | 2
  Pneumonia | 0 | 2
  High potassium | 0 | 1
  Hyperuricemia | 0 | 1
  Confusion | 0 | 1
  Dizziness | 0 | 1
  Speech impairment | 0 | 2
  Chest pain | 0 | 1
  Extremity pain | 0 | 2
  Muscle pain | 0 | 1
  Secondary malignancy - MDS | 0 | 1

3. Secondary Outcome: Cytostatic Overall Response Rate
Description: * Cytostatic overall response rate = CR + PR + SD greater than or equal to 6 months
  * Definitions per 2007 Cheson Lymphoma Response Criteria
Time Frame: From 6 months through 3.5 years after study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 42
Participants | 15 | 18

4. Secondary Outcome: Participant Response Rate in Relapsed or Refractory cHL.
Description: -Definitions per 2007 Cheson Lymphoma Response Criteria
Time Frame: Through 3.5 years from study entry or until disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 42
Participants
  CR | 1 | 3
  PR | 7 | 9
  SD | 13 | 11
  PD | 14 | 14
  Not evaluable | 3 | 4
  Unknown | 0 | 1

5. Secondary Outcome: Time to Progression (TTP).
Description: -Time to progression (TTP) is defined as the time from study entry until documented lymphoma progression or death as a result of lymphoma.
Time Frame: Through 3.5 years from study entry or until disease progression
Population: (2) participants were not evaluable in Cohort 2 because 2 patients did not have progression, death dates, or last follow-up dates so time to progression cannot be calculated.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2
Number analyzed (Participants) | 38 | 40
months | 3.68 [2 to 19] | 4.08 [2 to 24]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from entry onto the clinical trial until death as a result of any cause.
Time Frame: Through 3.5 years from study entry or until disease progression
Population: 1 participant was not evaluable in Cohort 1 and 5 participants were not evaluable in Cohort 2 because these participants did not have death dates or last follow-up dates so overall survival cannot be calculated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 37 | 37
months | 17.434 [13.355 to 30.493] | 23.717 [17.039 to NA] — There are too few deaths after this time point to define upper limit of the confidence interval unambiguously.

7. Secondary Outcome: Relapse Free Survival (RFS)
Time Frame: Through 3.5 years from study entry or until disease progression
Population: 2 participants in Cohort 2 were not evaluable because these patients did not have a date of progression, treatment failure, death or last follow-up so RFS could not be calculated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 40
months | 3.78 [1.84 to 6.45] | 3.93 [1.88 to 6.84]

8. Secondary Outcome: Event Free Survival (EFS).
Description: -Event-free survival (time to treatment failure) is measured from the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death).
Time Frame: Through 3.5 years from study entry or until disease progression
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 40
months | 3.78 [1.84 to 6.45] | 3.93 [1.88 to 6.84]

9. Secondary Outcome: Duration of Response
Description: -Duration of response: defined as the interval from the date of response (CR or PR) is documented to the date of progression, taking as reference the smallest measurements recorded since the treatment started
Time Frame: Through 3.5 years from study entry or until disease progression
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Number analyzed (Participants) | 38 | 40
months | 3.68 [2 to 19] | 4.08 [2 to 24]

ADVERSE EVENTS:
Arm/Group | Cohort 1 - Lenalidomide Daily on Days 1-21 | Cohort 2 - Lenalidomide Daily on Days 1-28
Serious Adverse Events (participants affected / at risk) | 9/38 | 10/42
Other Adverse Events (participants affected / at risk) | 38/38 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Lenalidomide Daily on Days 1-21 (N=38) | Cohort 2 - Lenalidomide Daily on Days 1-28 (N=42)
Infection with normal ANC (pneumonia) (Infections and infestations) | 1 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Febrile neutropenia (Infections and infestations) | 0 | 1
Leukopenia (Investigations) | 0 | 1
Secondary malignancy - MDS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Infection - lung (Infections and infestations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pregnancy (Reproductive system and breast disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Hearing loss (Ear and labyrinth disorders) | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General pain (General disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 1
Increased bilirubin (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Lenalidomide Daily on Days 1-21 (N=38) | Cohort 2 - Lenalidomide Daily on Days 1-28 (N=42)
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abscess (Skin and subcutaneous tissue disorders) | 0 | 1
Alkaline phosphatase (Investigations) | 11 | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Anorexia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (joint) (Musculoskeletal and connective tissue disorders) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Benign colon polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bilirubin (Investigations) | 5 | 7
Body aches (Musculoskeletal and connective tissue disorders) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Chest pain (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 6 | 4
Chills (General disorders) | 3 | 2
Conjuctivitis (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 13 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Creatinine (Investigations) | 6 | 5
Cutaneous horn, left arm (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 7
Diffuse body pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Disseminated cryptococcus (Infections and infestations) | 0 | 1
Distension/bloating (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 5
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (SOB) (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema (General disorders) | 5 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Esophagus pain (Gastrointestinal disorders) | 2 | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Facial numbness (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 19 | 18
Febrile neutropenia (Infections and infestations) | 1 | 1
Fever - no infection (General disorders) | 4 | 4
Flashing lights (Eye disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Flu-like syndrome (General disorders) | 5 | 0
Headache (Nervous system disorders) | 4 | 5
Hemoglobin (Blood and lymphatic system disorders) | 23 | 21
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
High calcium (Metabolism and nutrition disorders) | 2 | 2
High glucose (Metabolism and nutrition disorders) | 7 | 9
High magnesium (Metabolism and nutrition disorders) | 0 | 1
High potassium (Metabolism and nutrition disorders) | 3 | 2
High sodium (Metabolism and nutrition disorders) | 7 | 0
Hypertension (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 2 | 2
Infection with neutropenia (Infections and infestations) | 2 | 2
Infection with unknown ANC (Infections and infestations) | 0 | 1
Infection without neutropenia (Infections and infestations) | 12 | 9
Insomnia (Psychiatric disorders) | 0 | 1
Kidney stone (Renal and urinary disorders) | 0 | 1
Left ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukocytes (WBC) (Investigations) | 29 | 32
Liver dysfunction/failure (Hepatobiliary disorders) | 1 | 0
Loss of balance (Nervous system disorders) | 1 | 0
Low albumin (Metabolism and nutrition disorders) | 17 | 9
Low calcium (Metabolism and nutrition disorders) | 11 | 12
Low glucose (Metabolism and nutrition disorders) | 5 | 2
Low potassium (Metabolism and nutrition disorders) | 14 | 14
Low sodium (Metabolism and nutrition disorders) | 12 | 7
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0
Lymphopenia (Investigations) | 17 | 21
Memory impairment (Nervous system disorders) | 1 | 1
Mood alteration - Agitation (Psychiatric disorders) | 1 | 0
Mood alteration - Anxiety (Psychiatric disorders) | 1 | 1
Mood alteration - Depression (Psychiatric disorders) | 2 | 1
Mood alteration - NOS (Psychiatric disorders) | 1 | 1
Mucositis (Gastrointestinal disorders) | 3 | 2
Muscle pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 7
Nausea (Gastrointestinal disorders) | 14 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Neuropathic pain (Nervous system disorders) | 2 | 0
Neutrophils (ANC) (Investigations) | 25 | 28
Night sweats (Endocrine disorders) | 0 | 2
PTT (Investigations) | 0 | 1
Paleness (Skin and subcutaneous tissue disorders) | 0 | 1
Platelets (Investigations) | 21 | 26
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 13 | 6
SGOT (AST) (Investigations) | 10 | 8
SGPT (ALT) (Investigations) | 14 | 9
Schleraderma (Skin and subcutaneous tissue disorders) | 0 | 1
Sensory neuropathy (Nervous system disorders) | 8 | 4
Sinusitis (Infections and infestations) | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Sweating (General disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 0
Taste alteration (Gastrointestinal disorders) | 0 | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1
Thyroglossal duct cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor flare (General disorders) | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Voice changes (hoarseness) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 2
Watery eyes (Eye disorders) | 1 | 0
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 4 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes